CLINICAL TRIAL: NCT01316939
Title: A 52 Week Randomised, Double-blind, Placebo-controlled Study to Investigate the Efficacy and Safety of GSK1605786A in the Maintenance of Remission in Subjects With Crohn's Disease
Brief Title: GSK1605786A in the Maintenance of Remission in Subjects With Crohn's Disease
Acronym: SHIELD-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated due to the lack of efficacy of GSK1605786A in Crohn's disease based on the results of Study CCX114151.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 114157; 2010-022383-12 (EudraCT Number)
Record Dates: First submitted 2011-03-03; First posted 2011-03-16 (Estimated); Results first posted 2017-09-07 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-08

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease, oral CCR9 antagonist, placebo-controlled, maintenance of remission, 52-week treatment, quality of life
MeSH Terms: conditions — Crohn Disease | interventions — CCX282-B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- GSK1605786A once daily (Experimental): 500 milligrams once daily
  Interventions: Drug: GSK1605786A
- GSK1605786A twice daily (Experimental): 500 milligrams twice daily
  Interventions: Drug: GSK1605786A

INTERVENTIONS:
Drug: GSK1605786A — GSK1605786A 500 milligrams once daily
  Arms: GSK1605786A once daily
Drug: Placebo — Placebo
  Arms: Placebo
Drug: GSK1605786A — GSK1605786A 500 milligrams twice daily
  Arms: GSK1605786A twice daily

SUMMARY:
A randomised, double-blind, placebo-controlled study to evaluate the efficacy and safety of two doses (500 mg once daily and 500 mg twice daily) of GSK1605786A in maintaining remission over 52 weeks in adult subjects with Crohn's disease. Efficacy will be assessed by the Crohn's Disease Activity Index (CDAI) score. Eligible subjects will have achieved response (CDAI decrease of at least 100 points) and/or remission (CDAI less than 150) in a prior GSK sponsored induction study. The primary endpoint will be proportion of subjects in remission at both Weeks 28 and 52. Safety will be assessed by recording of adverse events, clinical laboratory parameters including liver function tests, vital signs and electrocardiogram. Population pharmacokinetics will evaluate the two doses of GSK1605786A. Health outcomes assessments will include changes in Inflammatory Bowel Disease Questionnaire (IBDQ), SF-36v2, EQ-5D, Work Productivity and Activity Impairment - Crohn's Disease (WPAI-CD) and disability.

DETAILED DESCRIPTION:
This is a multi-centre, randomised, placebo-controlled, double-blind parallel group study in adult subjects with Crohn's disease who previously achieved clinical response (CDAI decrease of at least 100 points) and/or remission (CDAI less than 150) in a prior Phase III induction study (Study CCX114151 or another GSK sponsored induction study). Subjects will be randomised to 52 weeks of oral treatment with GSK1605786A 500 mg once daily or 500 mg twice daily or placebo. Subjects who are receiving concomitant corticosteroids at entry will undergo dose tapering following a defined schedule. Subjects who complete the treatment period may be eligible to enter an open-label extension study. Subjects who experience disease worsening and require additional (rescue) treatment will be withdrawn and may be eligible to enter the open-label study. Subjects who do not enter the open-label study must complete a follow-up assessment 4 weeks after completion of treatment. Approximately 756 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Subjects achieving clinical response (CDAI decrease of at least 100 points) and/or remission (CDAI less than 150) upon completion of treatment in Study CCX114151 or another GSK sponsored induction study
* Written informed consent prior to any CCX114157 specific study procedures
* Females of child-bearing potential must be sexually inactive or commit to use of consistent and correct use of contraceptive methods with a failure rate of less than 1 percent
* Stable doses of Crohn's disease medications
* Subjects on corticosteroids at entry must be willing to undergo corticosteroid dose taper during the study

Exclusion Criteria:

* If female, is pregnant, has a positive pregnancy test or is breast-feeding
* Subjects with known or suspected coeliac disease or a positive screening test (anti-tissue transglutaminase antibodies) should have been excluded from enrolment into the induction studies. Subjects in whom a diagnosis of coeliac disease is subsequently suspected should have this excluded with testing for anti-tissue transglutaminase antibodies prior to enrolment into the maintenance study.
* Known or suspected fixed symptomatic small bowel stricture
* Enterocutaneous, abdominal or pelvic fistulae likely to require surgery during the study period
* Current sepsis or infections requiring intravenous antibiotic therapy for greater than 2 weeks
* Evidence of hepatic dysfunction, viral hepatitis, or liver function abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2011-05-09 (Actual); Primary Completion 2013-10-23 (Actual); Study Completion 2013-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (214):
- United States (51):
  - GSK Investigational Site, Little Rock, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Lakewood, Colorado
  - GSK Investigational Site, Littleton, Colorado
  - GSK Investigational Site, Hamden, Connecticut
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Port Orange, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Suwanee, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Hammond, Louisiana
  - GSK Investigational Site, Monroe, Louisiana
  - GSK Investigational Site, Chevy Chase, Maryland
  - GSK Investigational Site, Towson, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Chesterfield, Michigan
  - GSK Investigational Site, Troy, Michigan
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Lee's Summit, Missouri
  - GSK Investigational Site, Mexico, Missouri
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, East Setauket, New York
  - GSK Investigational Site, Great Neck, New York
  - GSK Investigational Site, Lake Success, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Germantown, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Ogden, Utah
  - GSK Investigational Site, Christiansburg, Virginia
  - GSK Investigational Site, Danville, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin
- Australia (8):
  - GSK Investigational Site, Bankstown, New South Wales
  - GSK Investigational Site, Hersten, Queensland
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Kurralta Park, South Australia
  - GSK Investigational Site, Box Hill, Victoria
  - GSK Investigational Site, Fitzroy, Victoria
  - GSK Investigational Site, Prahran, Victoria
  - GSK Investigational Site, Fremantle, Western Australia
- Austria (5):
  - GSK Investigational Site, Hall in Tirol
  - GSK Investigational Site, Linz
  - GSK Investigational Site, Oberpullendorf
  - GSK Investigational Site, St.Veit/Glan
  - GSK Investigational Site, Vienna
- Belgium (6):
  - GSK Investigational Site, Bonheiden
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Kortrijk
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Roeselare
- Bulgaria (3):
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Varna
- Canada (12):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Abbotsford, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
- GSK Investigational Site, Viña del Mar, Chile
- Czechia (4):
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Ostrava - Vitkovice
  - GSK Investigational Site, Prague
- Denmark (5):
  - GSK Investigational Site, Aalborg
  - GSK Investigational Site, Aarhus
  - GSK Investigational Site, Herlev
  - GSK Investigational Site, Hvidovre
  - GSK Investigational Site, Odense
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- France (8):
  - GSK Investigational Site, Clichy
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Saint-Priest-en-Jarez
  - GSK Investigational Site, Vandœuvre-lès-Nancy
- Germany (7):
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Brinkum/Stuhr, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Minden, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Hong Kong (2):
  - GSK Investigational Site, Hong Kong
  - GSK Investigational Site, Shatin, New Territories
- Hungary (6):
  - GSK Investigational Site, Békéscsaba
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Mosonmagyaróvár
  - GSK Investigational Site, Szekszárd
  - GSK Investigational Site, Vác
- Israel (10):
  - GSK Investigational Site, Afula
  - GSK Investigational Site, Beersheba
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Holon
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Ramat Gan
  - GSK Investigational Site, Tel Aviv
  - GSK Investigational Site, Ẕerifin
- Italy (4):
  - GSK Investigational Site, Palermo, Sicily
  - GSK Investigational Site, Genova
  - GSK Investigational Site, Modena
  - GSK Investigational Site, Roma
- Japan (10):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- Netherlands (4):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Ede
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Rotterdam
- New Zealand (4):
  - GSK Investigational Site, Dunedin
  - GSK Investigational Site, Lower Hutt
  - GSK Investigational Site, Otahuhu, Auckland
  - GSK Investigational Site, Tauranga
- Norway (2):
  - GSK Investigational Site, Tromsø
  - GSK Investigational Site, Tønsberg
- Poland (5):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Sopot
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Wroclaw
- Portugal (3):
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Porto
  - GSK Investigational Site, Viseu
- Russia (9):
  - GSK Investigational Site, Irkutsk
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Lipetsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Rostov-on-Don
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Tomsk
- Slovakia (5):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Nitra
  - GSK Investigational Site, Nové Mesto nad Váhom
  - GSK Investigational Site, Prešov
  - GSK Investigational Site, Trnava
- South Africa (4):
  - GSK Investigational Site, Bellville
  - GSK Investigational Site, Claremont
  - GSK Investigational Site, Observatory
  - GSK Investigational Site, Parktown
- South Korea (4):
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Wŏnju
- Spain (8):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Elche
  - GSK Investigational Site, Fuenlabrada (Madrid)
  - GSK Investigational Site, Galdakao/Vizcaya
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marbella
  - GSK Investigational Site, Sabadell (Barcelona)
  - GSK Investigational Site, Santander (Cantabria)
- Sweden (2):
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Stockholm
- Switzerland (2):
  - GSK Investigational Site, Bern
  - GSK Investigational Site, Zurich
- GSK Investigational Site, Taichung, Taiwan
- GSK Investigational Site, Ankara, Turkey (Türkiye)
- Ukraine (8):
  - GSK Investigational Site, Chernivtsi
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Odesa
  - GSK Investigational Site, Simferopol
  - GSK Investigational Site, Vinnytsia
- United Kingdom (8):
  - GSK Investigational Site, Harrow, Middlesex
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Edinburgh
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Oxford
  - GSK Investigational Site, Salford

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 128 centers in 28 countries with sites in North America, Europe, Israel, South Africa, Japan, Republic of Korea, Hong Kong, Australia, and New Zealand from 09 May 2011 and 23 October 2013.
Pre-assignment Details: The study was planned to randomize approximately 756 participants (252 participants per group) from induction studies CCX114151 and CCX114643. However a total of 229 participants (159 who participated in study CCX114151 and 70 who participated in study CCX114643) were randomized and comprised the analysis population for this study.
Groups:
- Placebo: Eligible participants received 52 weeks randomized, double-blind treatment with oral matching placebo capsules to GSK1605786A 500 milligram (mg) capsules.
- GSK1605786A 500 mg Once Daily: Eligible participants received 52 weeks randomized, double-blind treatment with oral GSK1605786A 500 mg capsules once daily.
- GSK1605786A 500 mg BID: Eligible participants received 52 weeks randomized, double-blind treatment with oral GSK1605786A 500 mg capsules twice daily (BID).
Period: Overall Study
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID
Started | 76 | 77 | 76
Completed | 13 | 9 | 7
Not Completed | 63 | 68 | 69
Not completed — Study closed/terminated | 26 | 25 | 23
Not completed — Lack of Efficacy | 24 | 25 | 25
Not completed — Adverse Event | 9 | 12 | 11
Not completed — Withdrawal by Subject | 1 | 3 | 6
Not completed — Physician Decision | 2 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Met Liver chemistry stopping criteria | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Eligible participants received 52 weeks randomized, double-blind treatment with oral matching placebo capsules to GSK1605786A 500 mg capsules.
- GSK1605786A 500 mg BID: Eligible participants received 52 weeks randomized, double-blind treatment with oral GSK1605786A 500 mg capsules BID.
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID | Total
Number analyzed (Participants) | 76 | 77 | 76 | 229
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.2 (13.20) | 36.7 (13.00) | 38.8 (12.75) | 37.9 (12.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 35 | 42 | 123
  Male | 30 | 42 | 34 | 106
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 4 | 7 | 6 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 3
  White | 70 | 67 | 69 | 206
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Clinical Remission (Crohn's Disease Activity Index , CDAI Score <150 Points) at Both Weeks 28 and 52 of the 52-week Treatment Period
Description: Clinical remission is defined as a CDAI score <150 points. In the missing=no effect imputation, participants with missing CDAI scores was considered not to be in clinical remission. Data for percentage of participants in at both Weeks 28 and 52 of the 52-week treatment period have been presented.
Time Frame: Week 28 and 52
Population: The Intent-to-Treat (ITT) Population comprised of all participants randomized to treatment who achieved a clinical response (CDAI decrease from baseline of >=100 points) or achieved clinical remission (CDAI <150 points).
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID
Number analyzed (Participants) | 76 | 77 | 76
Percentage of Participants | 10.5 | 6.5 | 3.9
Statistical Analysis 1: Comparison: Placebo vs GSK1605786A 500 mg Once Daily; Placebo Vs GSK1605786A 500 mg once daily at Week 28 and 52; Test type: Superiority or Other; Percent difference of participants = -4.0, 95% CI 2-sided [-12.9 to 4.8]
Statistical Analysis 2: Comparison: Placebo vs GSK1605786A 500 mg BID; Placebo Vs GSK1605786A 500 mg BID at Week 28 and 52; Test type: Superiority or Other; Percent difference of participants = -6.6, 95% CI 2-sided [-14.8 to 1.6]

2. Secondary Outcome: Percentage of Participants in Clinical Remission (CDAI Score <150 Points) and Not Taking Corticosteroids at Both Weeks 28 and 52 of the 52-week Treatment Period
Description: Clinical remission is defined as a CDAI score <150 points. A participant was considered to be not taking corticosteroids at Weeks 28 and 52 if the participant had not taken a corticosteroid for the 8 days prior to and the day of the CDAI assessment for each of Weeks 28 and 52. In the missing=no effect imputation, participants with missing CDAI scores was considered not to be in clinical remission. Data for percentage of participants in clinical remission and not taking corticosteroids at both Weeks 28 and 52 of the 52-week treatment period have been presented.
Time Frame: Week 28 and 52
Population: ITT Population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID
Number analyzed (Participants) | 76 | 77 | 76
Percentage of Participants | 9.2 | 5.2 | 3.9
Statistical Analysis 1: Comparison: Placebo vs GSK1605786A 500 mg Once Daily; Placebo Vs GSK1605786A 500 mg once daily at Week 28 and 52; Test type: Superiority or Other; Percent difference of participants = -4.0, 95% CI 2-sided [-12.2 to 4.2]
Statistical Analysis 2: Comparison: Placebo vs GSK1605786A 500 mg BID; Test type: Superiority or Other; Percent difference of participants = -5.3, 95% CI 2-sided [-13.1 to 2.6]

3. Secondary Outcome: Percentage of Participants in Clinical Remission at Both Weeks 28 and 52 of the 52-week Treatment Period Among Those Participants Who Were in Clinical Remission at Baseline
Description: Clinical remission is defined as a CDAI score <150 points. Among participants in remission at baseline, the percentage of participants with clinical remission at both Weeks 28 and 52 of the treatment period using the no effect imputation for missing data were to be compared between each GSK1605786A dose group and placebo using Fisher's exact test. Participants with missing CDAI scores were to be considered not to be in remission according to the missing=no effect imputation. The limited data resulting from early termination of Study CCX114157 did not allow any conclusions to be drawn about the efficacy of GSK1605786A in the maintenance of clinical remission in participants with Crohn's disease.
Time Frame: Week 28 and 52
Population: ITT Population. Following early termination of study CCX114157 data for Percentage of participants in clinical remission at both Weeks 28 and 52 of the 52-week treatment period among those participants who were in clinical remission at Baseline was not collected.
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Percentage of Participants in Clinical Remission at All Visits (Continuous Clinical Remission) During the 52-week Treatment Period Among Participants in Clinical Remission at Baseline
Description: The percentage of participants with clinical remission at all visits during the 52-week treatment period were to be summarized by treatment group for the subset of participants in remission at baseline, using the no effect imputation for missing data. Participants with missing CDAI scores were to be considered not to be in remission according to the missing=no effect imputation. Comparisons between each GSK1605786A dose group and placebo were to be made using Fisher's exact test.The limited data resulting from early termination of Study CCX114157 did not allow any conclusions to be drawn about the efficacy of GSK1605786A in the maintenance of clinical remission in participants with Crohn's disease.
Time Frame: Upto Week 52
Population: ITT Population. Following early termination of study CCX114157 data for Percentage of participants in clinical remission at all visits (continuous clinical remission) during the 52-week treatment period among participants in clinical remission at Baseline was not collected.
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants in Clinical Remission at Week 52
Description: The limited data resulting from early termination of Study CCX114157 did not allow any conclusions to be drawn about the efficacy of GSK1605786A in the maintenance of clinical remission in participants with Crohn's disease.
Time Frame: Week 52
Population: ITT Population. Following early termination of study CCX114157 data for Percentage of participants in clinical remission at Week 52 was not collected.
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants With a Clinical Response (CDAI Decrease >=100 Points) at Both Weeks 28 and 52 of the 52-week Treatment Period
Description: Clinical response is defined as a reduction from the induction study baseline CDAI score of >=100 points. The percentage of participants with a clinical response at both Weeks 28 and 52 of the 52-week maintenance treatment period in the ITT population using the no effect imputation for missing data were to be compared between each GSK1605786A dose group and placebo using Fisher's exact test. Participants with missing CDAI scores were to be considered non-responders according to the missing=no effect imputation. The limited data resulting from early termination of Study CCX114157 did not allow any conclusions to be drawn about the efficacy of GSK1605786A in the maintenance of clinical remission in participants with Crohn's disease.
Time Frame: Week 28 and 52
Population: ITT Population. Following early termination of study CCX114157 data for Percentage of participants with a clinical response (CDAI decrease >=100 points) at both Weeks 28 and 52 of the 52-week treatment period was not collected.
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Time to Induction of Clinical Remission in Participants Who Had Achieved Clinical Response During Induction Therapy But Were Not in Clinical Remission at Baseline
Description: The duration of time participants maintained clinical remission during the 52-week treatment period was to be defined as the time between Week 0 and the first visit where remission was not observed in those participants in remission at baseline. These time periods were to be summarized by treatment group using quartiles and their corresponding confidence intervals. Comparisons between each GSK1605786A dose group and placebo were to be made using log-rank tests. The limited data resulting from early termination of Study CCX114157 did not allow any conclusions to be drawn about the efficacy of GSK1605786A in the maintenance of clinical remission in participants with Crohn's disease.
Time Frame: Upto Week 52
Population: ITT Population. Following early termination of study CCX114157 data for Time to induction of clinical remission in participants who had achieved clinical response during induction therapy but were not in clinical remission at Baseline was not collected.
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline in CDAI Score at Weeks 4, 8, 12, 20, 28, 36, 44, and 52
Description: The CDAI score is used to quantify the symptoms of participants with Crohn's Disease. A score of 150 or below indicates remission and a score above 450 indicates extremely severe disease. A decrease in CDAI over time indicates improvement in disease activity. CDAI scores and changes in CDAI scores during the 52-week treatment period were to be summarized by treatment group at Weeks 4, 8, 12, 20, 28, 36, 44, and 52. The limited data resulting from early termination of Study CCX114157 did not allow any conclusions to be drawn about the efficacy of GSK1605786A in the maintenance of clinical remission in participants with Crohn's disease. Baseline was defined as value at Week 0. Change from Baseline was calculated by subtracting the Baseline value from the post-randomization value at the time of assessment.
Time Frame: Baseline (Week 0) and Weeks 4, 8, 12, 20, 28, 36, 44, and 52
Population: ITT Population. Following early termination of study CCX114157 data for Change from Baseline in CDAI score at Weeks 4, 8, 12, 20, 28, 36, 44, and 52 was not collected.
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score at Week 52
Description: The IBDQ consists of a self-administered 32-item questionnaire that evaluates quality of life across 4 dimensional scores: Bowel, Systemic, Social and Emotional. The IBDQ questionnaire was to be completed by each participant at baseline and at Weeks 28, and 52. The response to each question can range from 1 to 7, with 1 indicating severe problem and 7 indicating normal health. The total IBDQ is computed as the sum of the responses to the individual IBDQ questions. The total score can range between 32 to 224 with higher scores indicating a better quality of life. The limited data resulting from early termination of Study CCX114157 did not allow any conclusions to be drawn about the efficacy of GSK1605786A in the maintenance of clinical remission in participants with Crohn's disease. Baseline was defined as value at Week 0. Change from Baseline was calculated by subtracting the Baseline value from the post-randomization value at the time of assessment.
Time Frame: Baseline (Week 0) and Week 52
Population: ITT Population. Following early termination of study CCX114157 data for Change from Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) total score at Week 52 was not collected.
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, may jeopardize the participant or require medical or surgical intervention to prevent one of the other outcomes listed in the definition above, or is an event of possible drug-induced liver injury.
Time Frame: Upto 56 weeks
Population: The Safety Population comprised of all participants in the ITT population except those who did not take at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID
Number analyzed (Participants) | 76 | 77 | 76
Participants
  Any AE | 55 | 50 | 54
  Any SAE | 1 | 3 | 2

11. Secondary Outcome: Change From Baseline in Vital Sign Systolic Blood Pressure Systolic (SBP) and Diastolic Blood Pressure (DBP) Upto Week 56
Description: Vital sign assessments included SBP and DBP collected in supine position following 5 minutes of rest. Assessments were carried out at Weeks 4, 8, 12, 20, 28, 36, 44, 52 and Week 56. Baseline was defined as value at Week 0. Change from Baseline was calculated by subtracting the Baseline value from the post-randomization value at the time of assessment.
Time Frame: Baseline (Week 0) and Weeks 4, 8, 12, 20, 28, 36, 44, 52, 56
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID
Number analyzed (Participants) | 76 | 77 | 76
Millimeters of mercury
  SBP at Week 4: number analyzed (Participants) | 74 | 75 | 74
  SBP at Week 4 | -1.6 (13.08) | -0.9 (10.15) | 1.2 (11.06)
  SBP at Week 8: number analyzed (Participants) | 61 | 61 | 61
  SBP at Week 8 | -2.7 (13.75) | 0.7 (12.17) | 0.5 (12.91)
  SBP at Week 12: number analyzed (Participants) | 55 | 48 | 48
  SBP at Week 12 | -0.9 (11.93) | 0.9 (11.31) | 1.1 (13.53)
  SBP at Week 20: number analyzed (Participants) | 44 | 39 | 37
  SBP at Week 20 | -3.0 (12.70) | -0.7 (10.52) | 2.0 (9.64)
  SBP at Week 28: number analyzed (Participants) | 33 | 25 | 24
  SBP at Week 28 | 2.2 (10.62) | 1.2 (10.47) | 4.6 (11.63)
  SBP at Week 36: number analyzed (Participants) | 24 | 21 | 13
  SBP at Week 36 | 0.7 (13.50) | 2.1 (9.49) | 1.8 (15.76)
  SBP at Week 44: number analyzed (Participants) | 19 | 14 | 10
  SBP at Week 44 | -0.1 (12.59) | -1.6 (13.35) | 0.0 (13.18)
  SBP at Week 52: number analyzed (Participants) | 15 | 9 | 7
  SBP at Week 52 | -1.6 (13.80) | 1.0 (9.29) | 2.3 (13.25)
  SBP at Week 56: number analyzed (Participants) | 33 | 29 | 27
  SBP at Week 56 | -0.5 (13.19) | -1.3 (11.21) | 2.0 (11.09)
  DBP at Week 4: number analyzed (Participants) | 74 | 75 | 74
  DBP at Week 4 | -2.0 (9.90) | -2.0 (9.54) | -0.1 (9.05)
  DBP at Week 8: number analyzed (Participants) | 61 | 61 | 61
  DBP at Week 8 | -0.1 (10.39) | -0.6 (8.78) | -1.3 (8.03)
  DBP at Week 12: number analyzed (Participants) | 55 | 48 | 48
  DBP at Week 12 | -0.4 (10.22) | -1.5 (6.68) | -0.8 (10.12)
  DBP at Week 20: number analyzed (Participants) | 44 | 39 | 37
  DBP at Week 20 | -1.1 (9.33) | -2.0 (8.31) | 0.1 (8.17)
  DBP at Week 28: number analyzed (Participants) | 33 | 25 | 24
  DBP at Week 28 | 2.4 (8.00) | -1.2 (10.05) | 2.0 (6.13)
  DBP at Week 36: number analyzed (Participants) | 24 | 21 | 13
  DBP at Week 36 | -0.2 (9.94) | -0.5 (10.01) | 0.8 (9.04)
  DBP at Week 44: number analyzed (Participants) | 19 | 14 | 10
  DBP at Week 44 | 0.1 (12.09) | -3.0 (7.91) | -0.1 (10.29)
  DBP at Week 52: number analyzed (Participants) | 15 | 9 | 7
  DBP at Week 52 | -0.7 (8.99) | -1.4 (8.40) | 2.4 (8.00)
  DBP at Week 56: number analyzed (Participants) | 33 | 29 | 27
  DBP at Week 56 | 0.2 (9.05) | 0.1 (7.12) | 1.3 (9.53)

12. Secondary Outcome: Change From Baseline in Vital Sign Heart Rate Upto Week 56
Description: Vital sign assessment included heart rate collected in supine position following 5 minutes of rest. Assessments were carried out at Weeks 4, 8, 12, 20, 28, 36, 44, 52 and 56. Baseline was defined as value at Week 0. Change from Baseline was calculated by subtracting the Baseline value from the post-randomization value at the time of assessment.
Time Frame: Baseline (Week 0) and Weeks 4, 8, 12, 20, 28, 36, 44, 52 and 56
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID
Number analyzed (Participants) | 76 | 77 | 76
beats per minute
  Heart rate at Week 4: number analyzed (Participants) | 73 | 74 | 74
  Heart rate at Week 4 | 1.8 (11.06) | -2.2 (11.96) | 0.0 (10.17)
  Heart rate at Week 8: number analyzed (Participants) | 61 | 61 | 61
  Heart rate at Week 8 | 0.9 (10.85) | -0.4 (12.23) | -0.2 (12.93)
  Heart rate at Week 12: number analyzed (Participants) | 54 | 48 | 48
  Heart rate at Week 12 | 0.9 (10.27) | -2.4 (11.25) | -0.5 (11.24)
  Heart rate at Week 20: number analyzed (Participants) | 44 | 39 | 37
  Heart rate at Week 20 | -1.0 (9.59) | -0.8 (14.49) | -0.4 (13.83)
  Heart rate at Week 28: number analyzed (Participants) | 33 | 25 | 24
  Heart rate at Week 28 | 1.3 (11.65) | 0.5 (15.07) | -0.7 (11.56)
  Heart rate at Week 36: number analyzed (Participants) | 24 | 21 | 13
  Heart rate at Week 36 | -2.8 (9.92) | 2.4 (9.45) | 2.5 (8.11)
  Heart rate at Week 44: number analyzed (Participants) | 19 | 14 | 10
  Heart rate at Week 44 | 2.0 (10.96) | 2.6 (5.85) | 1.4 (11.22)
  Heart rate at Week 52: number analyzed (Participants) | 15 | 9 | 7
  Heart rate at Week 52 | 1.6 (8.87) | -0.1 (7.77) | 4.1 (8.55)
  Heart rate at Week 56: number analyzed (Participants) | 33 | 29 | 27
  Heart rate at Week 56 | -1.1 (8.79) | 1.5 (12.04) | -3.1 (8.43)

13. Secondary Outcome: Number of Participants With Shift From Baseline in Hematology Parameters
Description: Hematology parameters included platelets, neutrophils, lymphocytes, monocytes, eosinophils, basophils, hematocrit, red blood cell count, hemoglobin, white blood cell count and segmented neutrophils . Assessments were carried out at Weeks 4, 8, 12, 20, 28, 36, 44 and 52 and 56. The consolidated data for number of participants with shift from Baseline (change from Baseline) in hematology parameters characterized as high and low have been presented.
Time Frame: Upto Week 56
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID
Number analyzed (Participants) | 76 | 77 | 76
Participants
  Platelets low: number analyzed (Participants) | 76 | 76 | 75
  Platelets low | 1 | 1 | 0
  Platelets high: number analyzed (Participants) | 64 | 61 | 68
  Platelets high | 6 | 12 | 14
  Neutrophils low: number analyzed (Participants) | 76 | 76 | 74
  Neutrophils low | 3 | 2 | 1
  Neutrophils high: number analyzed (Participants) | 49 | 47 | 51
  Neutrophils high | 22 | 20 | 20
  Lymphocytes low: number analyzed (Participants) | 51 | 49 | 50
  Lymphocytes low | 19 | 19 | 14
  Lymphocytes high: number analyzed (Participants) | 75 | 76 | 74
  Lymphocytes high | 3 | 2 | 2
  Monocytes high: number analyzed (Participants) | 73 | 75 | 73
  Monocytes high | 7 | 4 | 7
  Eosinophils high: number analyzed (Participants) | 74 | 76 | 75
  Eosinophils high | 3 | 7 | 2
  Basophil high: number analyzed (Participants) | 76 | 76 | 75
  Basophil high | 0 | 0 | 1
  Hematocrit low: number analyzed (Participants) | 49 | 43 | 51
  Hematocrit low | 13 | 10 | 11
  Hematocrit high: number analyzed (Participants) | 75 | 76 | 73
  Hematocrit high | 1 | 1 | 2
  Red blood cell count low: number analyzed (Participants) | 37 | 40 | 42
  Red blood cell count low | 8 | 6 | 9
  Red blood cell count high: number analyzed (Participants) | 54 | 55 | 53
  Red blood cell count high | 1 | 0 | 2
  Hemoglobin low: number analyzed (Participants) | 37 | 35 | 47
  Hemoglobin low | 15 | 13 | 11
  Hemoglobin high: number analyzed (Participants) | 75 | 76 | 75
  Hemoglobin high | 1 | 0 | 0
  White blood cell count low: number analyzed (Participants) | 71 | 75 | 71
  White blood cell count low | 4 | 5 | 7
  White blood cell count high: number analyzed (Participants) | 63 | 62 | 65
  White blood cell count high | 9 | 12 | 6
  Segmented neutrophils low: number analyzed (Participants) | 76 | 76 | 74
  Segmented neutrophils low | 3 | 2 | 1
  Segmented neutrophils high: number analyzed (Participants) | 49 | 47 | 51
  Segmented neutrophils high | 22 | 20 | 20

14. Secondary Outcome: Number of Participants With Shift From Baseline in Clinical Chemistry Parameters
Description: Clinical chemistry parameters included total protein, phosphorous, albumin, sodium, potassium, chloride, calcium, glucose, gamma glutamyl transferase, total bilirubin, direct bilirubin, alkaline phosphatase, alanine amino transferase, aspartate amino transferase, blood urea nitrogen (BUN)/Urea, creatinine, uric acid, lactate dehydrogenase, bicarbonate, cholesterol and creatinine kinase. Assessments were carried out at Weeks 4, 8, 12, 20, 28, 36, 44, 52 and 56. The consolidated data for number of participants with shift from Baseline (change from Baseline) in clinical chemistry parameters characterized as high and low have been presented.
Time Frame: Upto Week 56
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID
Number analyzed (Participants) | 76 | 77 | 76
Participants
  Total protein low: number analyzed (Participants) | 73 | 71 | 68
  Total protein low | 3 | 7 | 5
  Total protein high: number analyzed (Participants) | 76 | 75 | 75
  Total protein high | 0 | 1 | 0
  Phosphorous low: number analyzed (Participants) | 69 | 74 | 73
  Phosphorous low | 2 | 9 | 13
  Phosphorous high: number analyzed (Participants) | 76 | 72 | 73
  Phosphorous high | 8 | 3 | 3
  Albumin low: number analyzed (Participants) | 75 | 71 | 74
  Albumin low | 1 | 2 | 3
  Albumin high: number analyzed (Participants) | 75 | 75 | 73
  Albumin high | 4 | 4 | 1
  Sodium low: number analyzed (Participants) | 74 | 75 | 73
  Sodium low | 1 | 1 | 3
  Sodium high: number analyzed (Participants) | 76 | 75 | 74
  Sodium high | 0 | 1 | 0
  Potassium low: number analyzed (Participants) | 76 | 73 | 75
  Potassium low | 4 | 1 | 4
  Potassium high: number analyzed (Participants) | 76 | 75 | 73
  Potassium high | 4 | 0 | 4
  Chloride low: number analyzed (Participants) | 76 | 75 | 75
  Chloride low | 0 | 0 | 1
  Chloride high: number analyzed (Participants) | 74 | 71 | 70
  Chloride high | 9 | 8 | 11
  Calcium low: number analyzed (Participants) | 72 | 72 | 71
  Calcium low | 3 | 5 | 7
  Calcium high: number analyzed (Participants) | 75 | 75 | 75
  Calcium high | 2 | 2 | 3
  Glucose low: number analyzed (Participants) | 74 | 73 | 71
  Glucose low | 6 | 8 | 12
  Glucose high: number analyzed (Participants) | 70 | 69 | 73
  Glucose high | 13 | 16 | 10
  Gamma glutamyl transferase high: number analyzed (Participants) | 68 | 68 | 71
  Gamma glutamyl transferase high | 5 | 6 | 10
  Total bilirubin high: number analyzed (Participants) | 75 | 77 | 74
  Total bilirubin high | 4 | 3 | 2
  Direct bilirubin high: number analyzed (Participants) | 76 | 77 | 75
  Direct bilirubin high | 1 | 1 | 1
  Alkaline phosphatase high: number analyzed (Participants) | 75 | 76 | 74
  Alkaline phosphatase high | 8 | 4 | 7
  Alanine amino transferase high: number analyzed (Participants) | 74 | 77 | 74
  Alanine amino transferase high | 5 | 3 | 8
  Asparatate amino transferase high: number analyzed (Participants) | 74 | 76 | 76
  Asparatate amino transferase high | 9 | 2 | 5
  BUN/Urea low: number analyzed (Participants) | 71 | 71 | 68
  BUN/Urea low | 4 | 6 | 5
  BUN/Urea high: number analyzed (Participants) | 76 | 75 | 75
  BUN/Urea high | 1 | 0 | 2
  Creatinine low: number analyzed (Participants) | 65 | 63 | 59
  Creatinine low | 6 | 8 | 12
  Creatinine high: number analyzed (Participants) | 76 | 75 | 74
  Creatinine high | 1 | 0 | 0
  Uric acid low: number analyzed (Participants) | 74 | 72 | 69
  Uric acid low | 3 | 3 | 3
  Uric acid high: number analyzed (Participants) | 72 | 75 | 74
  Uric acid high | 0 | 1 | 4
  Bicarbonate low: number analyzed (Participants) | 70 | 70 | 67
  Bicarbonate low | 21 | 16 | 18
  Lactate dehydrogenase high: number analyzed (Participants) | 75 | 73 | 75
  Lactate dehydrogenase high | 1 | 1 | 1
  Cholesterol high: number analyzed (Participants) | 57 | 61 | 68
  Cholesterol high | 7 | 4 | 11
  Creatinine kinase high: number analyzed (Participants) | 74 | 73 | 74
  Creatinine kinase high | 7 | 4 | 8

15. Secondary Outcome: Change From Baseline in Liver Function Test Parameter Total Bilirubin at Weeks 2, 4, 6, 8, 10, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52 and 56.
Description: Liver function test parameter included total bilirubin. Assessments were carried out at Weeks 2, 4, 6, 8, 10, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52 and 56. Baseline was defined as value at Week 0. Change from Baseline was calculated by subtracting the Baseline value from the post-randomization value at the time of assessment.
Time Frame: Baseline (Week 0) and Weeks 2, 4, 6, 8, 10, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52 and 56.
Population: Safety Population. Only those participants available at the specified time points were analyzed
Measure: Mean (Standard Deviation); unit: micromoles per liter
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID
Number analyzed (Participants) | 76 | 77 | 76
micromoles per liter
  Week 2: number analyzed (Participants) | 74 | 75 | 74
  Week 2 | 0.7 (3.21) | 0.0 (2.09) | -0.7 (2.48)
  Week 4: number analyzed (Participants) | 71 | 67 | 71
  Week 4 | 0.7 (3.46) | 0.0 (2.33) | -0.1 (2.24)
  Week 6: number analyzed (Participants) | 64 | 61 | 63
  Week 6 | 0.9 (2.29) | 0.1 (2.60) | -0.4 (2.95)
  Week 8: number analyzed (Participants) | 61 | 56 | 57
  Week 8 | 1.0 (3.38) | 0.2 (2.49) | 0.0 (2.31)
  Week 10: number analyzed (Participants) | 56 | 49 | 51
  Week 10 | 0.9 (3.46) | 0.5 (3.25) | -0.1 (3.27)
  Week 12: number analyzed (Participants) | 61 | 45 | 48
  Week 12 | 0.8 (2.70) | 0.2 (2.42) | 0.6 (3.33)
  Week 16: number analyzed (Participants) | 48 | 41 | 42
  Week 16 | 0.8 (3.75) | 0.8 (2.99) | -0.2 (2.00)
  Week 20: number analyzed (Participants) | 43 | 36 | 36
  Week 20 | 1.4 (3.07) | 0.9 (3.25) | 0.4 (2.89)
  Week 24: number analyzed (Participants) | 37 | 32 | 29
  Week 24 | 1.0 (3.26) | 0.8 (2.63) | 0.8 (4.27)
  Week 28: number analyzed (Participants) | 31 | 26 | 23
  Week 28 | 0.8 (3.37) | 0.4 (2.08) | 0.2 (4.30)
  Week 32: number analyzed (Participants) | 26 | 23 | 19
  Week 32 | 0.5 (2.37) | 0.2 (2.41) | 0.8 (5.70)
  Week 36: number analyzed (Participants) | 23 | 19 | 13
  Week 36 | 0.4 (2.62) | 0.6 (3.09) | 0.5 (2.44)
  Week 40: number analyzed (Participants) | 23 | 15 | 10
  Week 40 | 0.7 (2.52) | -0.5 (2.67) | 0.7 (3.16)
  Week 44: number analyzed (Participants) | 18 | 14 | 9
  Week 44 | 1.4 (2.79) | 0.0 (1.66) | 1.0 (6.44)
  Week 48: number analyzed (Participants) | 14 | 11 | 8
  Week 48 | 1.0 (4.49) | -1.4 (3.35) | -1.5 (6.97)
  Week 52: number analyzed (Participants) | 14 | 9 | 7
  Week 52 | 0.7 (4.81) | 0.6 (1.42) | -1.7 (9.53)
  Week 56: number analyzed (Participants) | 33 | 31 | 28
  Week 56 | 0.2 (3.69) | 1.4 (2.81) | 1.8 (3.47)

16. Secondary Outcome: Change From Baseline in Liver Function Test Parameter Albumin at Weeks 2, 4, 6, 8, 10, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and 56
Description: Liver function test parameter included albumin. Assessments were carried out at Weeks 2, 4, 6, 8, 10, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and 56.Baseline was defined as value at Week 0. Change from Baseline was calculated by subtracting the Baseline value from the post-randomization value at the time of assessment.
Time Frame: Baseline (Week 0) and Weeks 2, 4, 6, 8, 10, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and 56
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID
Number analyzed (Participants) | 76 | 77 | 76
grams per liter
  Week 2: number analyzed (Participants) | 4 | 8 | 7
  Week 2 | -0.3 (1.26) | 0.0 (2.51) | -0.1 (1.35)
  Week 4: number analyzed (Participants) | 70 | 66 | 69
  Week 4 | 0.7 (2.20) | 0.1 (2.39) | -0.2 (2.30)
  Week 6: number analyzed (Participants) | 1 | 3 | 7
  Week 6 | -1.0 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | -1.0 (2.00) | -0.6 (2.30)
  Week 8: number analyzed (Participants) | 61 | 56 | 57
  Week 8 | 0.2 (2.44) | 0.3 (2.37) | -0.6 (2.63)
  Week 10: number analyzed (Participants) | 6 | 4 | 5
  Week 10 | -2.0 (2.97) | -1.5 (2.08) | -1.4 (1.34)
  Week 12: number analyzed (Participants) | 50 | 45 | 48
  Week 12 | 0.0 (2.48) | 0.0 (2.43) | 0.0 (2.70)
  Week 16: number analyzed (Participants) | 3 | 5 | 4
  Week 16 | -3.0 (2.65) | -1.0 (3.00) | -1.5 (2.52)
  Week 20: number analyzed (Participants) | 43 | 35 | 36
  Week 20 | 0.4 (2.02) | 0.7 (2.78) | 0.0 (2.42)
  Week 24: number analyzed (Participants) | 5 | 4 | 3
  Week 24 | -0.2 (4.55) | -2.3 (4.35) | -4.0 (3.61)
  Week 28: number analyzed (Participants) | 30 | 24 | 23
  Week 28 | 0.1 (2.06) | 0.1 (4.47) | 0.5 (2.89)
  Week 32: number analyzed (Participants) | 0 | 3 | 0
  Week 32 |  | -4.0 (4.36) |
  Week 36: number analyzed (Participants) | 23 | 19 | 13
  Week 36 | -0.2 (2.78) | 0.7 (4.01) | 0.4 (2.79)
  Week 40: number analyzed (Participants) | 2 | 0 | 0
  Week 40 | 0.5 (2.12) |  |
  Week 44: number analyzed (Participants) | 18 | 14 | 8
  Week 44 | -0.2 (2.55) | 0.0 (2.69) | 0.4 (2.33)
  Week 48: number analyzed (Participants) | 1 | 1 | 1
  Week 48 | 2.0 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 1.0 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 1.0 (NA) — Standard deviation could not be calculated as a single participant was analyzed.
  Week 52: number analyzed (Participants) | 14 | 9 | 7
  Week 52 | -0.1 (2.14) | -1.3 (1.94) | 1.9 (2.27)
  Week 56: number analyzed (Participants) | 33 | 31 | 26
  Week 56 | -1.0 (2.48) | -0.5 (3.52) | -0.2 (3.03)

17. Secondary Outcome: Change From Baseline in Liver Function Test Parameter Alanine Amino Transferase, Aspartate Amino Transferase, Alkaline Phosphatase and Gamma Glutamyl Transferase at Weeks 2, 4, 6, 8, 10, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and 56
Description: Liver function test parameters included alanine amino transferase, aspartate amino transferase, alkaline phosphatase and gamma glutamyl transferase. Assessments were carried out at Weeks 2, 4, 6, 8, 10, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and 56. Baseline was defined as value at Week 0. Change from Baseline was calculated by subtracting the Baseline value from the post-randomization value at the time of assessment.
Time Frame: Baseline (Week 0) and Weeks 2, 4, 6, 8, 10, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and 56
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: units per liter
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID
Number analyzed (Participants) | 76 | 77 | 76
units per liter
  Alanine amino transferase at Week 2: number analyzed (Participants) | 74 | 75 | 74
  Alanine amino transferase at Week 2 | -1.0 (14.70) | 0.3 (5.88) | 0.2 (6.27)
  Alanine amino transferase at Week 4: number analyzed (Participants) | 71 | 67 | 71
  Alanine amino transferase at Week 4 | 0.2 (8.93) | -0.6 (4.83) | -0.1 (6.94)
  Alanine amino transferase at Week 6: number analyzed (Participants) | 64 | 61 | 63
  Alanine amino transferase at Week 6 | 0.4 (11.92) | 1.1 (6.66) | 0.3 (7.35)
  Alanine amino transferase at Week 8: number analyzed (Participants) | 61 | 56 | 57
  Alanine amino transferase at Week 8 | 0.0 (9.46) | -0.2 (6.20) | 1.0 (6.43)
  Alanine amino transferase at Week 10: number analyzed (Participants) | 56 | 49 | 51
  Alanine amino transferase at Week 10 | -2.1 (8.15) | -0.5 (5.24) | 0.9 (7.33)
  Alanine amino transferase at Week 12: number analyzed (Participants) | 51 | 45 | 48
  Alanine amino transferase at Week 12 | -2.7 (8.60) | -0.6 (5.13) | 0.6 (7.40)
  Alanine amino transferase at Week 16: number analyzed (Participants) | 48 | 41 | 42
  Alanine amino transferase at Week 16 | -1.4 (9.00) | 0.5 (7.69) | 0.4 (4.98)
  Alanine amino transferase at Week 20: number analyzed (Participants) | 43 | 36 | 36
  Alanine amino transferase at Week 20 | -2.7 (8.85) | -0.4 (7.07) | 1.4 (4.59)
  Alanine amino transferase at Week 24: number analyzed (Participants) | 37 | 32 | 29
  Alanine amino transferase at Week 24 | -1.3 (9.94) | -0.2 (6.25) | 2.3 (6.19)
  Alanine amino transferase at Week 28: number analyzed (Participants) | 31 | 26 | 23
  Alanine amino transferase at Week 28 | -1.6 (10.08) | -0.2 (5.91) | 0.3 (5.12)
  Alanine amino transferase at Week 32: number analyzed (Participants) | 26 | 23 | 19
  Alanine amino transferase at Week 32 | -2.3 (9.48) | -0.8 (6.81) | 11.1 (35.32)
  Alanine amino transferase at Week 36: number analyzed (Participants) | 23 | 19 | 13
  Alanine amino transferase at Week 36 | -2.3 (8.17) | -0.6 (7.46) | 5.4 (10.74)
  Alanine amino transferase at Week 40: number analyzed (Participants) | 23 | 15 | 10
  Alanine amino transferase at Week 40 | -3.4 (10.74) | 0.1 (10.24) | 6.0 (10.13)
  Alanine amino transferase at Week 44: number analyzed (Participants) | 18 | 14 | 9
  Alanine amino transferase at Week 44 | -3.2 (13.37) | -1.5 (7.72) | 0.3 (4.82)
  Alanine amino transferase at Week 48: number analyzed (Participants) | 14 | 11 | 8
  Alanine amino transferase at Week 48 | -3.8 (13.98) | -2.0 (12.21) | -0.6 (6.52)
  Alanine amino transferase at Week 52: number analyzed (Participants) | 14 | 9 | 7
  Alanine amino transferase at Week 52 | -5.1 (11.47) | -1.2 (11.41) | -1.3 (5.22)
  Alanine amino transferase at Week 56: number analyzed (Participants) | 33 | 31 | 28
  Alanine amino transferase at Week 56 | -5.8 (28.79) | 0.4 (8.11) | 10.3 (41.19)
  Aspartate amino transferase at Week 2: number analyzed (Participants) | 74 | 75 | 74
  Aspartate amino transferase at Week 2 | 0.4 (12.18) | 0.3 (3.76) | 0.6 (5.41)
  Aspartate amino transferase at Week 4: number analyzed (Participants) | 71 | 67 | 71
  Aspartate amino transferase at Week 4 | 0.5 (7.19) | 0.1 (4.24) | -0.2 (5.45)
  Aspartate amino transferase at Week 6: number analyzed (Participants) | 64 | 61 | 63
  Aspartate amino transferase at Week 6 | 1.2 (9.18) | 0.8 (3.99) | -0.1 (3.94)
  Aspartate amino transferase at Week 8: number analyzed (Participants) | 61 | 56 | 57
  Aspartate amino transferase at Week 8 | 0.1 (6.39) | 0.0 (4.07) | 1.0 (4.58)
  Aspartate amino transferase at Week 10: number analyzed (Participants) | 56 | 49 | 50
  Aspartate amino transferase at Week 10 | -0.7 (5.17) | 0.6 (3.94) | 0.8 (4.18)
  Aspartate amino transferase at Week 12: number analyzed (Participants) | 51 | 45 | 48
  Aspartate amino transferase at Week 12 | 0.4 (8.38) | 0.5 (5.97) | 1.1 (6.11)
  Aspartate amino transferase at Week 16: number analyzed (Participants) | 48 | 41 | 32
  Aspartate amino transferase at Week 16 | 0.0 (7.57) | 1.5 (5.29) | 0.4 (4.24)
  Aspartate amino transferase at Week 20: number analyzed (Participants) | 43 | 36 | 36
  Aspartate amino transferase at Week 20 | -0.2 (7.18) | 0.8 (4.74) | 0.2 (5.02)
  Aspartate amino transferase at Week 24: number analyzed (Participants) | 37 | 32 | 29
  Aspartate amino transferase at Week 24 | 0.0 (8.35) | 0.2 (4.52) | 1.7 (6.21)
  Aspartate amino transferase at Week 28: number analyzed (Participants) | 31 | 26 | 23
  Aspartate amino transferase at Week 28 | 1.3 (10.01) | 0.5 (4.52) | -0.9 (4.42)
  Aspartate amino transferase at Week 32: number analyzed (Participants) | 26 | 23 | 19
  Aspartate amino transferase at Week 32 | -0.2 (7.06) | -0.6 (6.67) | 4.9 (17.50)
  Aspartate amino transferase at Week 36: number analyzed (Participants) | 22 | 19 | 13
  Aspartate amino transferase at Week 36 | 0.0 (8.17) | 0.3 (4.36) | 3.3 (7.00)
  Aspartate amino transferase at Week 40: number analyzed (Participants) | 23 | 15 | 10
  Aspartate amino transferase at Week 40 | -0.7 (9.95) | -0.5 (3.66) | 3.8 (8.43)
  Aspartate amino transferase at Week 44: number analyzed (Participants) | 18 | 14 | 9
  Aspartate amino transferase at Week 44 | -1.3 (7.14) | -0.8 (5.03) | -0.8 (4.09)
  Aspartate amino transferase at Week 48: number analyzed (Participants) | 14 | 11 | 8
  Aspartate amino transferase at Week 48 | -0.1 (11.65) | -3.4 (8.87) | -0.4 (6.32)
  Aspartate amino transferase at Week 52: number analyzed (Participants) | 14 | 9 | 7
  Aspartate amino transferase at Week 52 | -1.4 (10.05) | -0.9 (3.98) | -1.0 (2.83)
  Aspartate amino transferase at Week 56: number analyzed (Participants) | 33 | 31 | 28
  Aspartate amino transferase at Week 56 | -2.5 (17.99) | -0.3 (4.13) | 5.4 (20.70)
  Alkaline phosphatase at Week 2: number analyzed (Participants) | 74 | 75 | 74
  Alkaline phosphatase at Week 2 | -0.2 (7.42) | 1.3 (9.54) | 0.4 (9.96)
  Alkaline phosphatase at Week 4: number analyzed (Participants) | 71 | 67 | 71
  Alkaline phosphatase at Week 4 | 0.1 (9.30) | 2.0 (10.63) | 0.4 (11.00)
  Alkaline phosphatase at Week 6: number analyzed (Participants) | 64 | 61 | 63
  Alkaline phosphatase at Week 6 | 1.0 (11.21) | 3.6 (11.28) | 1.0 (11.16)
  Alkaline phosphatase at Week 8: number analyzed (Participants) | 61 | 56 | 57
  Alkaline phosphatase at Week 8 | 1.7 (12.04) | 3.9 (12.61) | 0.2 (11.21)
  Alkaline phosphatase at Week 10: number analyzed (Participants) | 56 | 49 | 51
  Alkaline phosphatase at Week 10 | -1.4 (10.54) | 5.6 (12.55) | 2.8 (12.93)
  Alkaline phosphatase at Week 12: number analyzed (Participants) | 51 | 45 | 48
  Alkaline phosphatase at Week 12 | 1.2 (10.99) | 5.6 (14.85) | 2.4 (11.38)
  Alkaline phosphatase at Week 16: number analyzed (Participants) | 48 | 41 | 42
  Alkaline phosphatase at Week 16 | 1.5 (13.71) | 7.2 (13.16) | 3.4 (13.23)
  Alkaline phosphatase at Week 20: number analyzed (Participants) | 43 | 36 | 36
  Alkaline phosphatase at Week 20 | 3.7 (13.70) | 9.3 (16.74) | 2.0 (12.80)
  Alkaline phosphatase at Week 24: number analyzed (Participants) | 37 | 32 | 29
  Alkaline phosphatase at Week 24 | 1.9 (13.77) | 9.2 (17.74) | 3.4 (11.00)
  Alkaline phosphatase at Week 28: number analyzed (Participants) | 31 | 26 | 23
  Alkaline phosphatase at Week 28 | 1.9 (16.62) | 12.2 (16.71) | -0.6 (12.53)
  Alkaline phosphatase at Week 32: number analyzed (Participants) | 26 | 23 | 19
  Alkaline phosphatase at Week 32 | -1.0 (16.55) | 10.5 (19.52) | 4.3 (9.63)
  Alkaline phosphatase at Week 36: number analyzed (Participants) | 23 | 19 | 13
  Alkaline phosphatase at Week 36 | 2.3 (18.43) | 9.4 (16.98) | 6.3 (13.11)
  Alkaline phosphatase at Week 40: number analyzed (Participants) | 23 | 15 | 10
  Alkaline phosphatase at Week 40 | 1.5 (18.60) | 6.5 (6.71) | -0.2 (9.14)
  Alkaline phosphatase at Week 44: number analyzed (Participants) | 18 | 14 | 9
  Alkaline phosphatase at Week 44 | 2.6 (17.32) | 6.0 (9.88) | -3.6 (8.31)
  Alkaline phosphatase at Week 48: number analyzed (Participants) | 14 | 11 | 8
  Alkaline phosphatase at Week 48 | 10.6 (23.54) | 1.1 (19.93) | -5.5 (11.25)
  Alkaline phosphatase at Week 52: number analyzed (Participants) | 14 | 9 | 7
  Alkaline phosphatase at Week 52 | 2.1 (13.76) | 3.9 (10.28) | 3.9 (9.58)
  Alkaline phosphatase at Week 56: number analyzed (Participants) | 33 | 31 | 28
  Alkaline phosphatase at Week 56 | 3.5 (12.84) | 3.8 (14.98) | 4.9 (8.29)
  Gamma glutamyl transferase at Week 2: number analyzed (Participants) | 74 | 75 | 74
  Gamma glutamyl transferase at Week 2 | -3.0 (8.06) | 1.8 (13.22) | 0.4 (8.89)
  Gamma glutamyl transferase at Week 4: number analyzed (Participants) | 71 | 67 | 71
  Gamma glutamyl transferase at Week 4 | -4.2 (9.86) | -0.4 (12.58) | 2.1 (11.32)
  Gamma glutamyl transferase at Week 6: number analyzed (Participants) | 64 | 61 | 63
  Gamma glutamyl transferase at Week 6 | -5.0 (15.47) | 1.7 (13.10) | 1.9 (10.50)
  Gamma glutamyl transferase at Week 8: number analyzed (Participants) | 61 | 56 | 57
  Gamma glutamyl transferase at Week 8 | -1.2 (24.86) | 1.1 (16.05) | 2.0 (7.55)
  Gamma glutamyl transferase at Week 10: number analyzed (Participants) | 56 | 49 | 51
  Gamma glutamyl transferase at Week 10 | -6.2 (11.03) | 0.7 (14.38) | 2.2 (6.71)
  Gamma glutamyl transferase at Week 12: number analyzed (Participants) | 51 | 45 | 48
  Gamma glutamyl transferase at Week 12 | -8.2 (15.00) | 0.5 (14.94) | 2.3 (8.21)
  Gamma glutamyl transferase at Week 16: number analyzed (Participants) | 48 | 41 | 42
  Gamma glutamyl transferase at Week 16 | -3.4 (19.57) | -0.9 (12.17) | 3.7 (8.72)
  Gamma glutamyl transferase at Week 20: number analyzed (Participants) | 43 | 36 | 36
  Gamma glutamyl transferase at Week 20 | -6.5 (17.94) | -1.9 (11.95) | 2.9 (8.57)
  Gamma glutamyl transferase at Week 24: number analyzed (Participants) | 37 | 32 | 29
  Gamma glutamyl transferase at Week 24 | -6.4 (15.11) | -3.0 (19.17) | 2.6 (7.95)
  Gamma glutamyl transferase at Week 28: number analyzed (Participants) | 31 | 26 | 23
  Gamma glutamyl transferase at Week 28 | -7.8 (25.33) | -4.3 (17.17) | 1.3 (6.56)
  Gamma glutamyl transferase at Week 32: number analyzed (Participants) | 26 | 23 | 19
  Gamma glutamyl transferase at Week 32 | -13.2 (31.99) | -9.0 (31.31) | 6.5 (13.53)
  Gamma glutamyl transferase at Week 36: number analyzed (Participants) | 23 | 19 | 13
  Gamma glutamyl transferase at Week 36 | -9.0 (27.65) | -6.7 (18.39) | 11.0 (13.38)
  Gamma glutamyl transferase at Week 40: number analyzed (Participants) | 23 | 15 | 10
  Gamma glutamyl transferase at Week 40 | -11.7 (21.56) | -6.1 (18.98) | 8.9 (10.49)
  Gamma glutamyl transferase at Week 44: number analyzed (Participants) | 18 | 14 | 9
  Gamma glutamyl transferase at Week 44 | -7.4 (15.82) | -8.6 (20.03) | 4.4 (9.15)
  Gamma glutamyl transferase at Week 48: number analyzed (Participants) | 14 | 11 | 8
  Gamma glutamyl transferase at Week 48 | -4.4 (9.80) | -13.5 (40.87) | 4.1 (9.30)
  Gamma glutamyl transferase at Week 52: number analyzed (Participants) | 14 | 9 | 7
  Gamma glutamyl transferase at Week 52 | -10.4 (19.75) | 0.0 (11.64) | 8.3 (10.40)
  Gamma glutamyl transferase at Week 56: number analyzed (Participants) | 33 | 31 | 26
  Gamma glutamyl transferase at Week 56 | -4.2 (12.03) | -3.4 (13.50) | 0.8 (21.68)

18. Secondary Outcome: Number of Participants With 12 Lead Electocardiogram (ECG) Abnormalities at Week 28 and 52
Description: A 12 lead ECG was collected at Weeks 28 and 52. ECG abnormalities were characterized as abnormal-not clinically significant (A-NCS) and abnormal-clinically significant (A-CS). A-NCS data for Week 28 and 52 have been presented.
Time Frame: Week 28 and 52
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID
Number analyzed (Participants) | 76 | 77 | 76
Participants
  A-NCS, Week 28: number analyzed (Participants) | 32 | 23 | 24
  A-NCS, Week 28 | 5 | 7 | 4
  A-NCS, Week 52: number analyzed (Participants) | 14 | 8 | 7
  A-NCS, Week 52 | 2 | 0 | 1

19. Secondary Outcome: Change From Baseline in Short Form - 36 Version 2 (SF-36 v2) at Weeks 28 and 52
Description: The SF-36v2 health survey is a self-administered, generic, 36-item questionnaire designed to measure 8 domains of functional health status and well-being: physical functioning, role-physical, bodily pain, general health perceptions, vitality, social functioning, role-emotional, and mental health. Each domain is scored from 0 (poorer health) to 100 (better health). SF-36 v2 items are scored such that a higher score indicates a better health state and better functioning. Data for change from Baseline in SF-36 v2 at Weeks 28 and 52 was not collected following early termination of this study. Baseline was defined as value at Week 0. Change from Baseline was calculated by subtracting the Baseline value from the post-randomization value at the time of assessment.
Time Frame: Baseline (Week 0) and Weeks 28 and 52
Population: ITT Population. Following early termination of study CCX114157 data for change from Baseline in SF-36 v2 at Weeks 28 and 52 was not collected.
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID
Number analyzed (Participants) | 0 | 0 | 0

20. Secondary Outcome: Change From Baseline in European Quality of Life (EuroQol ) Five Dimensions Questionnaire (EQ-5D) at Weeks 28 and 52
Description: EQ-5D self-reported questionnaire is used to measure health-related quality of life by measuring 5 dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ-5D questionnaire includes a visual analog scale (VAS) which records participants self-rated health status on a graduated (0-100) scale with higher scores indicating higher Health-Related Quality of Life (HRQoL). Data for Change from Baseline in EuroQol five dimensions questionnaire (EQ-5D) at Weeks 28 and 52 was not collected following early termination of this study. Baseline was defined as value at Week 0. Change from Baseline was calculated by subtracting the Baseline value from the post-randomization value at the time of assessment.
Time Frame: Baseline (Week 0) and Weeks 28 and 52
Population: ITT Population. Following early termination of study CCX114157 data for Change from Baseline in European Quality of Life (EuroQol ) five dimensions questionnaire (EQ-5D) at Weeks 28 and 52 was not collected.
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID
Number analyzed (Participants) | 0 | 0 | 0

21. Secondary Outcome: Change From Baseline in Work Productivity & Activity Impairment - Crohn's Disease (WPAI-CD) at Weeks 28 and 52
Description: WPAI measures the effect of your CD on your ability to work and perform regular activities. 6-items assess impairment in work productivity and daily activity during the 7 days before the assessment. It measures the percentage of overall impairment in work productivity and daily activity due to CD. A WPAI score of 0% = no impairment and a score of 100% = total loss of work productivity or activity. An absolute change in WPAI score of 7% is considered the minimum clinically important difference (MCID). Data for change from Baseline in WPAI-CD at Weeks 28 and 52 was not collected following early termination of this study. Baseline was defined as value at Week 0. Change from Baseline was calculated by subtracting the Baseline value from the post-randomization value at the time of assessment.
Time Frame: Baseline (Week 0) and Weeks 28 and 52
Population: ITT Population. Following early termination of study CCX114157 data for Change from Baseline in Work productivity & activity impairment - Crohn's disease (WPAI-CD) at Weeks 28 and 52 was not collected.
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID
Number analyzed (Participants) | 0 | 0 | 0

22. Secondary Outcome: Receipt of Disability Benefits at Weeks 28 and 52
Description: Receipt of disability benefits (Yes/No) was to be recorded at Weeks 0, 28 and 52 and Early Withdrawal visit if applicable. Change from baseline in receipt of disability benefits was to be compared between participants in remission versus participants not in remission using a Wilcoxon rank sum test. Data for Receipt of disability benefits at Weeks 28 and 52 was not collected following early termination of this study.
Time Frame: Weeks 28 and 52
Population: ITT population. Following early termination of study CCX114157 data for Receipt of disability benefits at Weeks 28 and 52 was not collected.
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID
Number analyzed (Participants) | 0 | 0 | 0

23. Secondary Outcome: Change From Baseline in Health-related Resource Utilization at Weeks 28 and 52
Description: Healthcare related resource utilization was to include: Hospitalizations (all cause and Crohn's disease related), Length of stay, Surgical procedures (all cause and Crohn's disease related), Outpatient visits (all cause and Crohn's disease related ). The frequency of hospitalizations, surgical procedures and hospital out-patient visits were to be recorded at Weeks 28 and 52. The number and percentage of participants reporting all cause and Crohn's disease -related hospitalizations, surgeries, and hospital out-patient visits were to be summarized and compared between each GSK1605786A dose group and placebo using Fisher's exact test. Data for Change from Baseline in health-related resource utilization at Weeks 28 and 52 was not collected following early termination of this study. Baseline was defined as value at Week 0. Change from Baseline was calculated by subtracting the Baseline value from the post-randomization value at the time of assessment.
Time Frame: Baseline (Week 0) and Weeks 28 and 52
Population: ITT Population. Following early termination of study CCX114157 data for Change from Baseline in health-related resource utilization at Weeks 28 and 52 was not collected.
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID
Number analyzed (Participants) | 0 | 0 | 0

24. Secondary Outcome: Change From Baseline in C Reactive Protein (CRP) at Weeks 28 and 52
Description: C-reactive protein (CRP) at was to be assessed at Weeks 4, 8, 12, 20, 28, 36, 44, 52 visit if applicable. Data for Change from Baseline in C reactive protein (CRP) at Weeks 28 and 52 was not collected following early termination of this study. Baseline was defined as value at Week 0. Change from Baseline was calculated by subtracting the Baseline value from the post-randomization value at the time of assessment.
Time Frame: Baseline (Week 0 and Weeks 28 and 52
Population: ITT Population. Following early termination of study CCX114157 data for Change from Baseline in C reactive protein (CRP) at Weeks 28 and 52 was not collected.
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID
Number analyzed (Participants) | 0 | 0 | 0

25. Secondary Outcome: Change From Baseline in Faecal Calprotectin at Weeks 28 and 52
Description: Stool sample for faecal calprotectin were to be collected at Weeks 28 and 52 visit if applicable. Data for Change from baseline in faecal calprotectin at Weeks 28 and 52 was not collected following early termination of this study. Baseline was defined as value at Week 0. Change from Baseline was calculated by subtracting the Baseline value from the post-randomization value at the time of assessment.
Time Frame: Baseline (Week 0) and Weeks 28 and 52
Population: ITT Population. Following early termination of study CCX114157 data for Change from Baseline in faecal calprotectin at Weeks 28 and 52 was not collected.
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 56
Description: Safety population was used for analysis.
Groups:
- GSK1605786A 500 mg Once Daily: Eligible participants received 52 weeks randomized, double-blind treatment with oral GSK1605786A 500 milligram (mg) capsules once daily.
Arm/Group | Placebo | GSK1605786A 500 mg Once Daily | GSK1605786A 500 mg BID
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/77 | 0/76
Serious Adverse Events (participants affected / at risk) | 1/76 | 3/77 | 2/76
Other Adverse Events (participants affected / at risk) | 39/76 | 35/77 | 41/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=76) | GSK1605786A 500 mg Once Daily (N=77) | GSK1605786A 500 mg BID (N=76)
Lower respiratory tract infecion (Infections and infestations) | 0 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=76) | GSK1605786A 500 mg Once Daily (N=77) | GSK1605786A 500 mg BID (N=76)
Crohn's disease (Gastrointestinal disorders) | 13 | 12 | 10
Abdominal pain (Gastrointestinal disorders) | 10 | 5 | 9
Diarrhoea (Gastrointestinal disorders) | 8 | 3 | 3
Nausea (Gastrointestinal disorders) | 6 | 1 | 6
Vomiting (Gastrointestinal disorders) | 4 | 2 | 3
Toothache (Gastrointestinal disorders) | 3 | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 4 | 1
Nasopharyngitis (Infections and infestations) | 9 | 9 | 9
Influenza (Infections and infestations) | 1 | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 6 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 5
Headache (Nervous system disorders) | 6 | 3 | 9
Rash (Skin and subcutaneous tissue disorders) | 7 | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 4

LIMITATIONS AND CAVEATS:
The limited data resulting from early termination of Study CCX114157 did not allow any conclusions to be drawn about the efficacy of GSK1605786A in the maintenance of clinical remission in participants with Crohn's disease.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.